CLINICAL TRIAL: NCT05450406
Title: The Inland Norway Healthy Life Center Study
Acronym: INHLCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Trainome-031
Record Dates: First submitted 2022-06-28; First posted 2022-07-08 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Non-Communicable Chronic Diseases; Obesity; Insulin Resistance; Musculoskeletal Diseases; Psychological Disorder; Cardiovascular Diseases
MeSH Terms: conditions — Noncommunicable Diseases; Obesity; Insulin Resistance; Musculoskeletal Diseases; Mental Disorders; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Participants in the intervention group will receive 12-week follow-up from the Healthy Life Center
  Interventions: Other: Physical activity
- Control group (No Intervention): Participants in the intervention group will not receive follow-up from the Healthy Life Center

INTERVENTIONS:
Other: Physical activity — The participants will receive the possibility to attend weekly endurance, resistance and yoga exercise sessions administered by the Healthy Life Center. They will also receive personalized follow-up from the Healthy Life Center, and have the possibility to exercise at the local gym.
  Arms: Intervention group

SUMMARY:
Healthy Life Centers (Norwegian, 'Frisklivssentralen') is a municipal service in Norway that aims to promote both physical and mental health, as well as to limit the development of non-communicable diseases. Previous research has shown that receiving follow-up from Healthy Life Centers has led to higher levels of daily physical activity, in addition to improved self-reported health and quality of life among the participants. However, there is a lack of studies that have examined what kind of physiological health effects can be expected from participating in the Healthy Life Center's follow-up.

In this study, responses to the 12-week physical activity program of the Healthy Life Center will be compared with the responses in a negative control group that does not receive such follow-up. Both the intervention group and the reference group (the negative control group) will carry out the same tests and measurements before and after the 12 week period. The tests will include measurements of anthropometric variables (body height, body weight and waist circumference), body composition, arterial stiffness, resting blood pressure and blood variables (blood glucose, long-term blood glucose, blood lipid profile and inflammation markers), in addition to physical tests of mobility, balance, maximum aerobic capacity (maximal oxygen consumption) and maximum muscle strength. Questionnaires related to adherence to the Healthy Life Center follow-up, socio-demographic variables, eating and drinking habits, activity level, perceived physical fitness, motivation for exercise, and health-related quality of life will also be included.

ELIGIBILITY:
Intervention group

Inclusion Criteria:

* >18 years of age
* Receiving follow-up from the Healthy Life Center

Exclusion Criteria:

* In average >1 weekly exercise training session the last three months

Reference group

Inclusion Criteria:

* >18 years of age

Exclusion Criteria:

* In average >1 weekly exercise training session the last three months
* Receiving follow-up from the Healthy Life Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption (measured in mL/kg body mass/min) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period

SECONDARY OUTCOMES:
Balance, measured using the "single leg stance test" (measured in seconds) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Mobility, measured using the "sit-and-reach" and the "back stretch" test (measured in centimeters) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Fat mass (measured in kilograms) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Lean mass (measured in kilograms) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Bone mineral density ( measured in g/cm2) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Visceral fat (measured in grams) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Blood glucose levels (serum, fasted state) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Cholesterol and total triglyceride levels (serum, fasted state) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Resting blood pressure | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Systemic inflammation markers (levels of c-reactive protein, TNF-alpha, interleukin 6 and interleukin 8 in serum, fasted state) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Arterial stiffness | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Health-related quality of life (measured using the SF-36 questionnaire; scores from 0-100, where a higher score means a better outcome) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Body mass index | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Maximal muscle strength (measured in newtons produced during a leg press exercise) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Maximal muscle power (measured in watts produced during a leg press exercise) | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Waist circumference | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period

OTHER OUTCOMES:
Activity level | From before to after the 12-week intervention/control period
  Difference in change between the two study arms from before to after the 12-week intervention/control period
Adherence to the 12-week intervention (measured as the number of sessions the participant attended divided by the number of sessions prescribed) | During the 12-week intervention
  For the intervention group
Compliance to the 12-week intervention (measured as the number of sessions the participant conducted the session as prescribed divided by the number of total sessions) | During the 12-week intervention
  For the intervention group